CLINICAL TRIAL: NCT04450394
Title: A Phase 2, Parallel, Comparator-Controlled Trial to Evaluate the Safety and Efficacy of LY3209590 in Insulin-Naïve Patients With Type 2 Diabetes Mellitus
Brief Title: A Phase 2 Study of LY3209590 in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17056; I8H-MC-BDCL (Other: Eli Lilly and Company); 2019-003339-53 (EudraCT Number)
Record Dates: First submitted 2020-06-26; First posted 2020-06-29 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3209590 Algorithm 1 (Paper) (Experimental): Algorithm 1 is a paper-based algorithm where dose adjustments were manually determined by the investigator based on fasting glucose and hypoglycemia data. LY3209590 was provided in a 20 milligram (mg) vial of reconstitutable lyophilized powder. Participants received individualized LY3209590 loading dose based on the baseline median fasting glucose and body weight by subcutaneous (SC) injection on day 1 followed by weekly adjustments for the first 12 weeks, then every 4 weeks, of a 26-week treatment period, to achieve target fasting glucose of <=100 milligrams per deciliter (mg/dL).
  Interventions: Drug: LY3209590
- LY3209590 Algorithm 2 (Digital) (Experimental): Algorithm 2 is a computer-based algorithm to determine dose adjustments. LY3209590 was provided in a 20 mg vial of reconstitutable lyophilized powder. Participants received individualized LY3209590 loading dose based on the baseline median fasting glucose and body weight by SC injection on day 1 followed by weekly adjustments for the first 12 weeks, then every 4 weeks, of a 26-week treatment period, to achieve target fasting glucose of <=100 mg/dL.
  As per protocol amendment (d) approved on 28-Oct-2020, this arm was terminated during the early enrollment phase due to technical issues with data entry.
  Interventions: Drug: LY3209590
- Insulin Degludec (Active Comparator): Insulin degludec was provided as 100 units/milliliter (U/mL) in a prefilled pen. Participants received individually adjusted doses once daily by SC injection with a starting dose of 10 units, during the 26-week treatment period, to achieve target fasting blood glucose of <=100 mg/dL.
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: LY3209590 — Administered SC
  Arms: LY3209590 Algorithm 1 (Paper); LY3209590 Algorithm 2 (Digital)
Drug: Insulin Degludec — Administered SC
  Arms: Insulin Degludec

SUMMARY:
The reason for this study is to see if the study drug LY3209590 is safe and effective in participants with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have type 2 diabetes mellitus according to the World Health Organization (WHO) criteria treated with a stable dose of metformin in combination with a stable dose of Dipeptidyl Peptidase IV (DPPIV) inhibitor and/or a Sodium-glucose co-transporter-2 (SGLT2) inhibitor for at least 3 months prior to screening
* Participants must have a HbA1c value of 7.0% to 9.5%, inclusive
* Participants must have a body mass index (BMI) between 20 and 45 kilograms per meter squared (kg/m²), inclusive

Exclusion Criteria:

* Have type 1 diabetes mellitus or latent autoimmune diabetes
* Have any episodes of severe hypoglycemia and/or hypoglycemia unawareness within the 6 months prior to screening
* Have any of the following cardiovascular (CV) conditions: acute myocardial infarction, New York Heart Association Class III or IV heart failure, or cerebrovascular accident (stroke)
* Have acute or chronic hepatitis, or obvious clinical signs or symptoms of any other liver disease
* Have an estimated glomerular filtration rate (eGFR) <30 milliliters/minute/1.73 m²
* Have active or untreated cancer
* Are receiving chronic (>14 days) systemic glucocorticoid therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5hours, EST), Study Director — Eli Lilly and Company
Locations (64):
- United States (31):
  - Syed Research Consultants Llc, Sheffield, Alabama
  - National Research Institute - Huntington Park, Huntington Park, California
  - National Research Institute - Wilshire, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Encompass Clinical Research, Spring Valley, California
  - CMR of Greater New Haven, Waterbury, Connecticut
  - ALL Medical Research, LLC, Cooper City, Florida
  - Jellinger and Lerman, MD PA dba The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Rophe Adult and Pediatric Medicine, Union City, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Elite Clinical Trials, Rexburg, Idaho
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Sky Clin Resch - Quinn HC, Ridgeland, Mississippi
  - Lillestol Research LLC, Fargo, North Dakota
  - Intend Research, LLC, Norman, Oklahoma
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Holston Medical Group, Bristol, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - Juno Research, Houston, Texas
  - Juno Research - Gessner, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (11):
  - Centro Médico Viamonte, CABA, Buenos Aires
  - Investigaciones Medicas Imoba Srl, CABA, Buenos Aires
  - Fundacion Sanatorio Guemes, CABA, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Caba, Buenos Aires
  - CEDIC, CABA, Buenos Aires
  - Instituto Médico Catamarca, Rosario, Santa Fe Province
  - CEMEDIC, Buenos Aires
  - Asociación de Beneficencia Hospital Sirio Libanés, Buenos Aires
  - Instituto Centenario, Ciudad Autonoma de Buenos Aire
  - Cent Priva Especiali Médicas Ambulatorias Inve Clin CEMAIC, Córdoba
  - Clínica Mayo, San Miguel de Tucumán
- Germany (8):
  - Diabetes- und Stoffwechselpraxis Bochum, Bochum, North Rhine-Westphalia
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Institut für Diabetesforschung GmbH Münster, Münster, North Rhine-Westphalia
  - Practice Dr.med. Denger and Dr.med. Pfitzner, Friedrichsthal, Saarland
  - Private Practice - Dr. Christine Kosch, Pirna, Saxony
  - SMO.MD GmbH, Magdeburg, Saxony-Anhalt
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Diabeteszentrum Hamburg West, Hamburg
- Poland (11):
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - Instytut Diabetologii Sp. z o.o, Warsaw, Masovian Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek, Henryk Rudzki, Ruda Śląska, Silesian Voivodeship
  - Centrum Kliniczno-Badawcze, Elblag
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - Gabinety TERPA, Lublin
  - OMEDICA Medical Center, Poznan
  - Praktyka Lekarska, Poznan
  - Poradnia Chorob Metabolicznych, Wierzchosławice
  - NZOZ Regionalna Poradnia Diabetologiczna, Wroclaw
- Puerto Rico (3):
  - Research and Cardiovascular Corp., Ponce, PR
  - GCM Medical Group, PSC - Hato Rey Site, San Juan, PR
  - Centro Profesional de Endocrinologia del Este, Yabucoa, PR

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Bue-Valleskey JM, Kazda CM, Ma C, Chien J, Zhang Q, Chigutsa E, Landschulz W, Haupt A, Frias JP. Once-Weekly Basal Insulin Fc Demonstrated Similar Glycemic Control to Once-Daily Insulin Degludec in Insulin-Naive Patients With Type 2 Diabetes: A Phase 2 Randomized Control Trial. Diabetes Care. 2023 May 1;46(5):1060-1067. doi: 10.2337/dc22-2396. PMID 36944059
- See also: A Phase 2 Study of LY3209590 in Participants With Type 2 Diabetes Mellitus — https://trials.lillytrialguide.com/en-US/trial/6qyhRt87M4hnov8DyzZZhb

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initially designed as 3 arms: LY3209590 Algorithm 1 (Paper), LY3209590 Algorithm 2 (Digital), and Insulin Degludec. However, it was amended to terminate the "LY3209590 Algorithm 2 (Digital)" arm during early enrollment phase due to technical issues with data entry. Thus, this arm was excluded from the outcome measure analyses, but safety data was analysed and reported.
Groups:
- LY3209590 Algorithm 2 (Digital): Algorithm 2 is a computer-based algorithm to determine dose adjustments. LY3209590 was provided in a 20 mg vial of reconstitutable lyophilized powder. Participants received individualized LY3209590 loading dose based on the baseline median fasting glucose and body weight by SC injection on day 1 followed by weekly adjustments for the first 12 weeks, then every 4 weeks, of a 26-week treatment period, to achieve target fasting glucose of <=100 mg/dL.
Period: Overall Study
Arm/Group | LY3209590 Algorithm 1 (Paper) | Insulin Degludec | LY3209590 Algorithm 2 (Digital)
Started | 129 | 135 | 14
Received at Least One Dose of Study Drug | 129 | 135 | 14
Completed | 119 | 121 | 14
Not Completed | 10 | 14 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 9 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- LY3209590 Algorithm 1 (Paper): Algorithm 1 is a paper-based algorithm where dose adjustments were manually determined by the investigator based on fasting glucose and hypoglycemia data. LY3209590 was provided in a 20 mg vial of reconstitutable lyophilized powder. Participants received individualized LY3209590 loading dose based on the baseline median fasting glucose and body weight by SC injection on day 1 followed by weekly adjustments for the first 12 weeks, then every 4 weeks, of a 26-week treatment period, to achieve target fasting glucose of <=100 mg/dL.
- Insulin Degludec: Insulin degludec was provided as 100 U/mL in a prefilled pen. Participants received individually adjusted doses once daily by SC injection with a starting dose of 10 units, during the 26-week treatment period, to achieve target fasting blood glucose of <=100 mg/dL.
- Total: Total of all reporting groups
Arm/Group | LY3209590 Algorithm 1 (Paper) | Insulin Degludec | LY3209590 Algorithm 2 (Digital) | Total
Number analyzed (Participants) | 129 | 135 | 14 | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (9.9) | 59.4 (9.1) | 56.3 (8.8) | 58.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 9 | 126
  Male | 71 | 76 | 5 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 59 | 8 | 128
  Not Hispanic or Latino | 68 | 76 | 6 | 150
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 14 | 1 | 19
  White | 123 | 119 | 12 | 254
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 29 | 27 | 0 | 56
  Puerto Rico | 9 | 4 | 2 | 15
  United States | 53 | 61 | 12 | 126
  Poland | 20 | 22 | 0 | 42
  Germany | 18 | 21 | 0 | 39
Haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of haemoglobin A. It is measured to identify average blood glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.05 (0.77) | 7.95 (0.75) | 8.38 (0.83) | 8.02 (0.77)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of haemoglobin A. It is measured to identify average blood glucose concentration over prolonged periods of time. Least squares (LS) mean change from baseline was analysed by mixed model repeated measures (MMRM) model with treatment, country, Dipeptidyl peptidase IV (DPPIV) (yes/no), Sodium-glucose Cotransporter-2 (SGLT2) (yes/no), baseline body mass index (BMI) [<30, >=30]), visit, and treatment by visit interaction as fixed effects and the baseline HbA1c as a covariate.
Time Frame: Baseline, Week 26
Population: All participants randomized to either LY3209590 Algorithm 1 (Paper) or Insulin degludec, received at least one dose of study drug and had baseline, post-baseline HbA1c data prior to treatment discontinuation.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | LY3209590 Algorithm 1 (Paper) | Insulin Degludec
Number analyzed (Participants) | 127 | 130
Percentage of HbA1c | -1.20 (0.076) | -1.26 (0.075)
Statistical Analysis 1: Comparison: LY3209590 Algorithm 1 (Paper) vs Insulin Degludec; Test type: Non-Inferiority — The non-inferiority margin is 0.4%. Non-inferiority is achieved if the upper limit of the 90% Confidence Interval is below 0.4; LS Mean Difference = 0.06, 90% CI 2-sided [-0.11 to 0.24]

2. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Description: LS mean change from baseline was analysed by MMRM model with treatment, country, DPPIV (yes/no), SGLT2 (yes/no), baseline BMI [<30, >=30]), visit, and treatment by visit interaction as fixed effects and the baseline fasting serum glucose as a covariate.
Time Frame: Baseline, Week 26
Population: All participants randomized to either LY3209590 Algorithm 1 (Paper) or Insulin degludec, received at least one dose of study drug and had baseline, post-baseline fasting serum glucose data prior to treatment discontinuation.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY3209590 Algorithm 1 (Paper) | Insulin Degludec
Number analyzed (Participants) | 126 | 130
milligrams per deciliter (mg/dL) | -50.7 (2.81) | -58.7 (2.83)

3. Secondary Outcome: Rate of Documented Hypoglycemia
Description: Documented hypoglycemia is defined as any time a participant reports a self-monitoring blood glucose <54 mg/dL (3.0 millimole per liter (mmol/L)). Rate of documented hypoglycemia per year during defined period is calculated by the number of documented hypoglycemia events within the period divided by the number of days participant at risk within the period*365.25 days.
Time Frame: Baseline through Week 26
Population: All participants randomized to either LY3209590 Algorithm 1 (Paper) or Insulin degludec, received at least one dose of study drug.
Measure: Number; unit: Events per participant per year
Arm/Group | LY3209590 Algorithm 1 (Paper) | Insulin Degludec
Number analyzed (Participants) | 129 | 135
Events per participant per year | 0.21 | 0.15

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of LY3209590
Description: AUC of LY3209590 was calculated for individual participants using the participants' Week 26 LY3209590 dose amount and estimated clearance value.
Time Frame: Week 26
Population: All participants randomized to LY3209590 Algorithm 1 (Paper), received at least one dose of study drug and had evaluable PK data at week 26.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole*hour per Liter (nmol*hr/L)
Arm/Group | LY3209590 Algorithm 1 (Paper)
Number analyzed (Participants) | 110
Nanomole*hour per Liter (nmol*hr/L) | 5890 (66)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (up to 31 weeks)
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | LY3209590 Algorithm 1 (Paper) | Insulin Degludec | LY3209590 Algorithm 2 (Digital)
All-Cause Mortality (participants affected / at risk) | 0/129 | 1/135 | 0/14
Serious Adverse Events (participants affected / at risk) | 6/129 | 4/135 | 1/14
Other Adverse Events (participants affected / at risk) | 18/129 | 19/135 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY3209590 Algorithm 1 (Paper) (N=129) | Insulin Degludec (N=135) | LY3209590 Algorithm 2 (Digital) (N=14)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/71 (0) | 1/76 (1) | 0/5 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3209590 Algorithm 1 (Paper) (N=129) | Insulin Degludec (N=135) | LY3209590 Algorithm 2 (Digital) (N=14)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 7 (8) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 7 (7) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was initially designed as 3 arms: LY3209590 Algorithm 1 (Paper), LY3209590 Algorithm 2 (Digital), and Insulin Degludec. However, it was amended to terminate the "LY3209590 Algorithm 2 (Digital)" arm during early enrollment phase due to technical issues with data entry. Thus, this arm was excluded from the outcome measure analyses, but safety data was analysed and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT04450394/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT04450394/SAP_001.pdf